

Ysbyty Athrofaol Cymru University Hospital of Wales



IRAS ID: 238464 Study ID Number:

Patient Identification Number:

## PARTICIPANT RE- CONSENT FORM 1 [Version 2.0 30/01/18]

| Title of Study: | Measuring Phys | ical Activity Levels in Criti | cal Care: A F | easibility | Study |
|---|---|---|---|---|---|
| Name of Researc | cher: Mrs Laura | a Jones, Dr Harriet Shann | on | Please in | iitial box |
| [version 2.0] for | the above study | derstand the information solution. I have had the opportunited have had these answe | ty to conside | r | |
| | • • • | n is voluntary and that I ar<br>ason, without my medical | | | |
| 3. I understand that relevant sections of my medical notes and data collected<br>during the study, may be looked at by individuals from regulatory authorities,<br>University College London or from Cardiff and Vale UHB, where it is relevant<br>to my taking part in this research. I give permission for these individuals to<br>have access to my records. | | | | | |
| | | eted by the activPAL <sup>™</sup> devarant for the device on my leg w | | | |
| 5. I agree to take | part in the above | study. | | | |
| 6. I would like to receive a copy of the findings of the study: Yes No | | | | | |
| Name of patient | | <br>Date | Signature | | |
| Name of person to | aking consent | <br>Date | Signature | | |